CLINICAL TRIAL: NCT02288273
Title: A Randomized Double-blind, Parallel-group Study to Evaluate the Effect of BYDUREON Compared With Placebo on 24-hour Glucose Control in Metformin-treated Patients With Type 2 Diabetes
Brief Title: Study to Evaluate the Effect of BYDUREON on 24-hour Glucose Control in Metformin Treated Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5551L00006
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bydureon (Experimental): Once weekly injected exenatide
  Interventions: Drug: Bydureon
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bydureon — Once weekly injection of 2mg bydureon (extended release exenatide) for 10 weeks.
  Other Names: exenatide
  Arms: Bydureon
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-blind, Parallel-group Study to Evaluate the Effect of Bydureon Compared with Placebo on 24-hour Glucose Control in Metformin-treated Patients with Type 2 Diabetes.

DETAILED DESCRIPTION:
A Randomized, Double-blind, Parallel-group Study to Evaluate the Effect of Bydureon Compared with Placebo on 24-hour Glucose Control in 110 Metformin-treated Patients with Type 2 Diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (T2DM) treated with stable dose of metformin > or = to 1500mg/day as monotherapy for at least 8 weeks
* Hemoglobin A1c (HbA1c) 7% to 10% at screening
* Body mass index (BMI) < or = to 45 kg/m2

Exclusion Criteria:

* History of taking antihyperglycemic therapy other than metformin or metformin extended release (XR) during the 8 weeks prior to screening
* History of taking a dipeptidyl peptidase-4 (DPP-4) inhibitor or pramlintide during 12 weeks prior to screening
* History of potent, inhaled or intrapulmonary steroids 3 months prior to screening or during the study
* History of prescription or over the counter weight loss medication during 3 months prior to screening
* Previous exposure to exenatide or any glucagon-like peptide-1 (GLP-1) receptor agonist during 6 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Research Site, Anaheim, California
  - Research Site, Chino, California
  - Research Site, Los Angeles, California
  - Research Site, North Hollywood, California
  - Research Site, Santa Ana, California
  - Research Site, Spring Valley, California
  - Research Site, Tustin, California
  - Research Site, Walnut Creek, California
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Edina, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Franklin, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Corpus Christi, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burke, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Olympia, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 239 subjects were screened in order to randomize 117 subjects; however, 116 subjects were included in the modified intent to treat population, which consisted of all randomized patients who received at least one dose of randomized study drug.
Groups:
- Once Weekly (EQW) + Met: Bydureon EQW + Metformin XR 1500-2000 mg
- Placebo + Met: Placebo + Metformin 1500 + 2000 mg
Period: Overall Study
Arm/Group | Once Weekly (EQW) + Met | Placebo + Met
Started | 61 | 56
Completed | 53 | 48
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Population: 239 subjects were screened in order to randomize 117 subjects; however, 116 subjects were included in the modified intent to treat population, which consisted of all randomized patients who received at least one dose of randomized study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Once Weekly (EQW) + Met | Placebo + Met | Total
Number analyzed (Participants) | 60 | 56 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (10.63) | 56 (9.80) | 55.6 (10.21)
Gender [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hour Mean Weighted Glucose
Description: Change in 24-hour mean weighted glucose from baseline (Day -1/1) to Day 6 of Week 4 (Day 27/28) and to Day 6 of Week 10 (Day 69/70).
Time Frame: Day 27/28
Measure: Mean (Standard Deviation); unit: (mg/dL)
Units Other Than Participants: (mg/dL)
Groups:
- EQW + Met: Bydureon EQW + Metformin 1500-2000 mg
Arm/Group | EQW + Met | Placebo + Met
Number analyzed (Participants) | 60 | 56
Number analyzed ((mg/dL)) | 60 | 56
(mg/dL)
  Baseline (Day -1/1) | 185.7 (41.99) | 183.8 (42.59)
  Day 27/28 | 158.3 (35.72) | 176.9 (44.03)
  Change from Baseline to Day 27/28 | -26.0 (3.58) | -5.3 (3.85)
  Change from Baseline to Day 69/70 | -30.8 (4.54) | -3.0 (4.78)
Statistical Analysis 1: Comparison: EQW + Met vs Placebo + Met; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: Change in 24-hour Mean Weighted Glucose Between Day 1 of Week 10 (Day 64/65) and Day 6 of Week 10 (Day 69/70) Within Each EQW-treated Patient
Time Frame: Day 64/65
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | EQW + Met | Placebo + Met
Number analyzed (Participants) | 60 | 56
mg/dL | 5.2 (3.46) | -6.9 (3.68)

3. Secondary Outcome: Change From Baseline (Day1) to Day 70 and Day 22 in FPG
Time Frame: Day 22/Day70
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | EQW + Met | Placebo + Met
Number analyzed (Participants) | 60 | 56
mg/dL
  Baseline to Day 22 | -29.6 (4.85) | -1.9 (4.99)
  Baseline to Day 70 | -41.9 (5.21) | -5.0 (5.53)

4. Secondary Outcome: Change From Baseline (Day -1) to Day 64 and Day 22 in 2- Hour Mean Weighted PPG (After the Breakfast Meal)
Time Frame: Day 22 and Day 64
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | EQW + Met | Placebo + Met
Number analyzed (Participants) | 60 | 56
mg/dL
  Baseline to Day 22 | -32.1 (5.30) | -2.0 (5.51)
  Baseline to Day 64 | -44.4 (5.62) | -6.0 (6.12)

5. Secondary Outcome: Average of Change in 24-hour Mean Weighted Glucose From Baseline to Week 4 and Baseline to Week 10
Time Frame: Week 4 and Week 10
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | EQW + Met | Placebo + Met
Number analyzed (Participants) | 60 | 56
mg/dL
  Change in mean weighted glucose baseline to Week 4 | -4.5 (1.09) | -1.8 (1.13)
  Change in mean weighted glucose baseline - Week 10 | -6.3 (1.31) | 0.7 (1.36)
  Change in MAGE (mg/dL) from baseline to Week 4 | -8.2 (3.13) | -3.8 (3.25)
  Change in MAGE (mg/dL) from baseline to Week 10 | -15.2 (3.51) | 2.9 (3.62)

6. Secondary Outcome: Change in HbA1c From Baseline to Day 22 and Baseline to Day 70
Time Frame: Day 22 and Day 70
Measure: Least Squares Mean (Standard Error); unit: % Alc
Arm/Group | EQW + Met | Placebo + Met
Number analyzed (Participants) | 60 | 56
% Alc
  Change from baseline to Day 22 | -0.30 (0.045) | -0.10 (0.047)
  Change from baseline to Day 70 | -0.92 (0.102) | -0.20 (0.108)

7. Secondary Outcome: Average of Change in 24-hour Mean Weighted Glucose From Baseline to Week 4 and Baseline to Week 10
Time Frame: Week 4 and Week 10
Measure: Least Squares Mean (Standard Error); unit: % times patients had specific CGM/24-hr
Arm/Group | EQW + Met | Placebo + Met
Number analyzed (Participants) | 60 | 56
% times patients had specific CGM/24-hr
  Change in times(%): PG<70 baseline to Week 4 | 0.5 (0.19) | 0.2 (0.19)
  Change in times (%): PG <70 baseline to Week 10 | 0.5 (0.21) | 0.1 (0.21)
  Change in %: 70 </= PG </=180 baseline to week 4 | 15.8 (2.37) | 4.1 (2.46)
  Change in %: 70 </= PG </=180 baseline to week 10 | 21.4 (2.99) | 1.3 (3.09)
  Change in times (%): PG >180 baseline to Week 4 | -16.2 (2.37) | -4.3 (2.47)
  Change in times (%): PG >180 baseline to Week 10 | -22.0 (3.04) | -1.4 (3.14)

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | EQW + Met | Placebo + Met
Serious Adverse Events (participants affected / at risk) | 4/60 | 1/56
Other Adverse Events (participants affected / at risk) | 35/60 | 26/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQW + Met (N=60) | Placebo + Met (N=56)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Acute Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than .02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQW + Met (N=60) | Placebo + Met (N=56)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 3 (3) | 3 (3)
Injection site nodule (General disorders) | 6 (6) | 0 (0)
Edema peripheral (General disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 1 (1)
Amylase increased (Investigations) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Glycosuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution & PI agree they will not use or disclose and confidential information to third parties for a period of 10 years from receipt.